CLINICAL TRIAL: NCT02579434
Title: Evaluation and Validation of Endogenous Markers for the Assessment of CYP3A Activity in Korean Healthy Subjects Using Metabolomics
Acronym: CYP3A_basal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Joo-Youn Cho, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CYP3A_basal
Record Dates: First submitted 2014-12-23; First posted 2015-10-19 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Healthy Volunteers
Keywords: CYP3A

ARMS (4):
- Male young adults (Experimental): Arm 1: Male healthy volunteers aged from 20 to 45 years Midazolam (IV) on day 1
  Interventions: Drug: Midazolam I.V.
- Male elderly adults (Experimental): Arm 2: Male healthy volunteers aged over 45 years Midazolam (IV) on day 1
  Interventions: Drug: Midazolam I.V.
- Female elderly adults (Experimental): Arm 3: Female healthy volunteers aged over 45 years Midazolam (IV) on day 1
  Interventions: Drug: Midazolam I.V.
- Female young adults (Experimental): Arm 4: Female healthy volunteers aged 20 to 45 years Midazolam (IV) on day 1, Day 15
  Interventions: Drug: Midazolam I.V.

INTERVENTIONS:
Drug: Midazolam I.V. — Midazolam I.V. 1mg/ml

SUMMARY:
The study objective is to evaluate and validate of endogenous markers for the assessment of CYP3A activity in Korean healthy subjects using metabolomics.

In part 1, total 75 healthy subjects (males and females) will be enrolled. In part 2, total 25 healthy female subject aged 20-45 years will be enrolled. In both part A and B, subjects will be administered midazolam I.V. 1 mg.

ELIGIBILITY:
Inclusion Criteria:

* Age: Between 20 to 80 years of age, inclusive
* Weight: Between 45 to 95 kg, within 17 - 28 of Body Mass Index
* Subject who agree contraception during the study
* Subject who are reliable and willing to make themselves available during the study period, are willing to follow the study protocol, and give their written informed consent voluntarily

Exclusion Criteria:

* History of hypersensitive reaction to medication (midazolam, ketoconazole, rifampicin)
* History of significant clinical illness needs medical caution, including cardiovascular, immunologic, hematologic, neuropsychiatric, respiratory, gastrointestinal, hepatic, or renal disease or other chronic disease history or evidence of drug abuse
* A subject whose lab test results are abnormal A subject whose systolic blood pressure is over 140 mmHg or below 90 mmHg and diastolic blood pressure is over 100 mmHg or below 50 mmHg
* Presence or history of drug abuse or positive result in urine drug screening test
* Blood donation during 2 months or apheresis during 1 month before the study Use any prescriptive medication
* Use of alcohol over 21 units/weeks
* Smoker who smoke more than 10 cigarettes per day
* Participation in clinical trials of any drug within 60 days prior to the participation of the study
* Use of grapefruit juice within 1 week before first dose
* Use of caffeine drink within 3 days before first dose
* Subject pregnant or breast-feeding
* Judged to be inappropriate for the study by the investigator

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Area under the curve of midazolam (AUC12h) | Up to 12 hours after midazolam administration
  Pharmacokinetics of midazolam
Metabolic ratio of steroids | 12h-12h
  endogenous metabolite profiles such as steroid (6beta-hydroxy-cortisol/cortisol, 6beta-hydroxy-cortisone/cortisone)
Clearance (CL) of midazolam | Up to 12 hours after midazolam administration
  Pharmacokinetics of midazolam

CONTACTS AND LOCATIONS:
Locations (1):
- Jieon Lee, Seoul, South Korea